CLINICAL TRIAL: NCT01376869
Title: Investigation of the Acute Cognitive, Mood and Autonomic Effects of Hops in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: The New Zealand Institute of Plant and Food Research Ltd. (Other Government)
Responsible Party: Principal Investigator, Crystal Haskell, Research Fellow, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21AO1
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Mood Modulation; Modulation of Cognition
Keywords: Hops; Mood; Cognitive Function; Bioavailability; Satiety; Blood Pressure; Heart rate
MeSH Terms: interventions — ALPL protein, human; Silicon Dioxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 102mg extract 1 hops (Active Comparator): Equivalent to 0.5g dry weight
  Interventions: Dietary Supplement: Hops Extract
- 410mg extract 1 hops (Active Comparator): Equivalent to 2g dry weight
  Interventions: Dietary Supplement: Hops Extract
- 79mg extract 2 hops (Active Comparator): Equivalent to 0.5g dry weight
  Interventions: Dietary Supplement: Hops Extract
- 316mg extract 2 hops (Active Comparator): Equivalent to 2g dry weight
  Interventions: Dietary Supplement: Hops Extract
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo (silica)

INTERVENTIONS:
Dietary Supplement: Hops Extract — All 150 participants will complete 1 study visit; receiving either of the 4 hops doses or placebo (silica). Computer generated random numbers will be used to allocate treatments to participant identification numbers. Treatment will be administered in capsule form and in a double blind manner.
  Arms: 102mg extract 1 hops; 316mg extract 2 hops; 410mg extract 1 hops; 79mg extract 2 hops
Other: Placebo (silica) — All 150 participants will complete 1 study visit; receiving either of the 4 hops doses or placebo (silica). Computer generated random numbers were used to allocate treatments to participant identification numbers. Treatment will be administered in capsule form and in a double blind manner.
  Arms: Placebo

SUMMARY:
Hops have been used for many years for their supposed sedative and anxiety reducing properties and can be found in many natural remedies for stress, anxiety and sleeping that are already available to buy.

However, human trials investigating the effects of hops have so far been limited to the effects of the combination of hops and valerian in relation to sleep. Such studies have identified that a valerian-hops mixture can result in improved sleep but Valerian alone has no effect.

The current study aims to investigate the effect of hops alone in healthy human participants aged 18-35 years.

ELIGIBILITY:
Inclusion Criteria:

* Male/female,
* Healthy
* Age 18-35 years old
* Non smoker
* Proficient in English
* Not taking any herbal or prescription medications
* Not pregnant seeking to become pregnant or breastfeeding

Exclusion Criteria:

* Allergy or hypersensitivity to any of the ingredients contained in the investigational product or any other foodstuff.
* Vegetarian (as the capsules contain gelatine).
* Have a history of neurological, vascular or psychiatric illness (including depressive illness and anxiety).
* Have a current/ history of drug or alcohol abuse.
* Currently take medication (excluding the contraceptive pill).
* High Blood Pressure (>140/90)
* BMI outside of the range 18- 34.9

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mood | across 3 hours
  * Mood as assessed by STAI, Bond-Lader mood scales, POMS, DEQ and stress/euphoria/sedation visual analogue scales (VAS).
  * The shift in mood (STAI, Bond-Lader, POMS, DEQ, Stress/Euphoria/Sedation VAS) inculcated by completion of cognitive tasks.
  * Heart rate and blood pressure.
  * The modulation of blood pressure and heart rate inculcated by completion of cognitive tasks.

SECONDARY OUTCOMES:
Satiety | across 3 hours
  * Satiety as assessed by VAS (hungry/full/desire to eat/food intake).
  * The modulation of satiety (VAS) inculcated by completion of the cognitive tasks.
Bioavailability of Hops | across 3 hours
  • Plasma hops levels are to be examined to assess bioavailability.
Cognition | across 3 hours
  * Performance on working memory tasks (2-back and logical reasoning).
  * Performance on serial subtraction element of a dual task.
  * Performance on word and picture recognition tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell, Study Director — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom